CLINICAL TRIAL: NCT02600650
Title: EndogenousTestosterone Response to a Testosterone Boosting Supplement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Canadian Memorial Chiropractic College (Other)
Collaborators: Iovate Health Sciences International Inc (Industry)
Responsible Party: Principal Investigator, Brian Budgell, Professor, Canadian Memorial Chiropractic College
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 151004
Record Dates: First submitted 2015-08-19; First posted 2015-11-09 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-11

CONDITIONS: Testosterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Receive daily authentic Testosterone boosting supplement
  Interventions: Dietary Supplement: Testosterone boosting supplement
- Placebo (Placebo Comparator): Receive daily placebo supplementation
  Interventions: Dietary Supplement: Placebo Comparator

INTERVENTIONS:
Dietary Supplement: Testosterone boosting supplement — Proprietary formulation of Testosterone boosting supplement administered daily
  Arms: Experimental
Dietary Supplement: Placebo Comparator — Daily administration of Placebo Comparator
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether a proprietary 'testosterone-boosting' supplement, when used as recommended by the manufacturer, results in an increase in testosterone levels as measured by a salivary free testosterone assay.

DETAILED DESCRIPTION:
The experimental intervention in this study is the daily administration of a testosterone boosting supplement or sham supplement for 4 weeks. The supplement will be administered daily in capsule form. The control group will be given a sham capsule containing the carrier components of the supplement. Participants will be asked not to modify their current lifestyle. Salivary testosterone levels will be assessed prior to the intervention to collect a baseline measurement for each subject, and following the intervention to evaluate any changes in hormone levels.

ELIGIBILITY:
Inclusion Criteria:

* Adult male aged 20 to 40 years.
* Fluent in English.

Exclusion Criteria:

* Currently receiving hormonal therapy or testosterone boosting supplement.
* Has received hormonal therapy or testosterone boosting supplement within 3 months prior to study.
* Has experienced adverse event following previous exposure to testosterone boosting supplements.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Change in concentration of salivary free testosterone from baseline measured by ELISA | 4 weeks
  Change in concentration of salivary free testosterone from baseline to 4 weeks will be measured by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: brian budgell, Ph.D., Principal Investigator — Canadian Memorial Chiropractic College
Locations (1):
- Canadian Memorial Chiropractic College, Toronto, Ontario, Canada